CLINICAL TRIAL: NCT03614442
Title: Evaluation of the Effect of Slopped Shoulder Implant Neck Versus Conventional Implant Neck Design on the Crestal Bone Level in the Maxilla: Randomized Clinical Trial (RCT)
Brief Title: Effect of Slopped Shoulder Implant Neck vs Conventional Implant Neck Design on Crestal Bone Level in the Maxilla
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hosam Ahmed Sharawi Shehabeldin, B.Sc. in Oral and Dental Medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: platform switching 2018
Record Dates: First submitted 2018-07-16; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-07

CONDITIONS: Missing Tooth
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: the design of the dental implant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- slopped shoulder implant (Experimental): The osteotomy site will be prepared using appropriate drill sizes with flapless approach, The implant (conventional neck implant design )will be inserted till the platform will be flushed with the crestal bone, The primary stability will be checked using torque wrench
  Interventions: Other: slopped shoulder implant
- conventional implant with flat platform (Active Comparator): inserted implant will be bone leveled implant (crestal maxi z) implant (conventional implant with platform). The primary stability will be checked using torque wrench
  Interventions: Other: slopped shoulder implant

INTERVENTIONS:
Other: slopped shoulder implant — different implant design to enhance soft and hard tissue outcome

SUMMARY:
In implant dentistry, platform switching is a method used to preserve alveolar bone levels around dental implants. The concept refers to using an implant with slopped shoulder neck of narrower diameter on implants of wider diameter, rather than placing abutments of similar diameter, referred to as platform matching.The aim of the study is to compare the effect of bone-level implants versus the conventional implant on oral soft tissues.

DETAILED DESCRIPTION:
Implant prosthesis allows normal muscle function, and the implant stimulates the bone and maintains its dimensions in a manner similar to healthy natural teeth. Crestal bone loss can result in increased bacterial accumulation resulting in secondary peri-implant inflammation and bone loss which can further result in loss of alveolar support, which in turn can lead to occlusal overload resulting in implant failure. In implant dentistry, platform switching is a method used to preserve alveolar bone levels around dental implants. The concept refers to using an implant with slopped shoulder neck of narrower diameter on implants of wider diameter, rather than placing abutments of similar diameter, referred to as platform matching. The authors developed the concept of slopped shoulder implant which results in an inward bone creeping at the coronal part of the implant to be in continuity with the alveolar bone crest.

The rational to use this type of implant allows an increase at residual crestal bone volume around the implant neck and has 3 merits:

1. Reduced mechanical stress at the implant neck area;
2. Repositioning of gingival papillae on the beveled neck implant (that is the physiologic condition);
3. proper vascular supply to the implant investing structure and bone tissue also because of reduced inter-implant space.

The aim of the study is to compare the effect of bone-level implants versus the conventional implant on oral soft tissues

ELIGIBILITY:
Inclusion Criteria:

* Good oral hygiene
* Systemically healthy (free from any systemic diseases).
* Adequate native bone to achieve implant primary stability
* Have had the tooth extraction at least 3 months before implant surgery.
* Did not receive soft or hard tissue augmentation before or in conjunction with implant surgery

Exclusion Criteria:

* Smokers
* Pregnant woman
* Had a history of alcoholism or drug abuse within the past 5 years.
* Had bruxism or clenching habits.
* Patients who refused to join the study.
* Had significant untreated periodontal disease or history of treated periodontitis.
* Had caries on teeth adjacent to the prospective implant site.
* Periapical infection.
* localized radiation therapy of the oral cavity; antitumor chemotherapy.
* poor oral hygiene

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2018-07-30 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
pink esthetic score(PES) | 8 months
  soft tissue esthetics scale : Seven variables will be evaluated vs. a natural reference tooth: mesial papilla, distal papilla, soft-tissue level, soft-tissue contour, alveolar process deficiency, soft-tissue color and texture. Using a 0-1-2 scoring system, 0 being the lowest, 2 being the highest value, the maximum achievable PES is 14.

SECONDARY OUTCOMES:
crestal bone resorption | 8 months
  bone loss around implant neck will be measured using (CBCT) cone beam computed tomography. On CBCT scans, the amount of bone resorption in the buccal, lingual/palatal, mesial and distal surfaces will be determined by measuring the distance from the platform of the implant to the alveolar crest (normal group: 0-1.5mm, mild bone loss: 1.6-3mm, moderate bone loss: 3.1-4.5mm and severe bone loss: >4.5mm)
implant stability | 8 months
  osteointegration of dental implant using (periotest device ).Periotest value range:
  * 8.0 to0.0 Good osseointegration
    * 0.1 to +9.9 the implant can be loaded
    * 10.0 or higher loading of the implant might or might not be possible

IPD SHARING:
Plan to Share IPD: Undecided